CLINICAL TRIAL: NCT04687774
Title: Real World Study of Exalt D Single-use Duodenoscope in ERCP Procedures in China
Brief Title: Exalt D Single-use Duodenoscope in ERCP Procedures in China
Acronym: ExaltDScope
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Strategy Adjustment
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: E7164
Record Dates: First submitted 2020-12-09; First posted 2020-12-29 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Cholangiopancreatography
Keywords: ERCP

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- single-arm study (Experimental): A single-arm of 30 treated patients is appropriate to generate additional local data on Exalt D Single-use Duodenoscope, since there is existing information in the previous study of Exalt D Single-use Duodenoscope in ERCP procedures and clinical literature regarding its performance.
  Interventions: Device: ExaltTM Model D Single-Use Duodenoscope

INTERVENTIONS:
Device: ExaltTM Model D Single-Use Duodenoscope — The Exalt™ Model D Single-Use Duodenoscope is a sterile, single-use endoscope that facilitates access to the duodenum, delivery of accessories, and live video when connected to an Exalt™ Controller.
  Other Names: ExaltTM Controller

SUMMARY:
Study Objective(s)：This study is to evaluate the feasibility, preliminary safety and performance of Exalt D Single-use Duodenoscope in ERCP procedures in China, to generate local real world data from a Chinese ERCP population.

Study Design：Prospective, single-arm study Planned Number of Subjects：Up to 35 to satisfy 30 treated cohort Primary Endpoint：Ability to complete the ERCP procedure for the intended indication(s) without crossing to reusable duodenoscope.

It is also considered as Exalt D's ability if the clinical effect is the same per the investigator's judgement in case of an endoscope change (non-Exalt D).

DETAILED DESCRIPTION:
Device Description：The Exalt™ Model D Single-Use Duodenoscope is a sterile, single-use endoscope that facilitates access to the duodenum, delivery of accessories, and live video when connected to an Exalt™ Controller.

The Exalt™ Controller is an electronic device that:

* Receives video signals from a Boston Scientific single-use endoscope,
* Processes the video signals,
* Outputs video images to a video monitor, and
* Outputs electrical signal(s) that interface with external image capture systems.

Study Design：This is a prospective, single-arm study with up to 35 subjects to satisfy 30 treated cohort in up to 3 centers. The study duration is expected to be approximately 7 months, assuming 6 months enrollment and 1 month follow up. The study duration for each subject is expected to be approximately 30 days.

Data Analyses：All statistical analyses will be done using The SAS System software, version 8 or higher (Copyright © 2000 SAS Institute Inc., SAS Campus Drive, Cary, North Carolina 27513, USA. All rights reserved).

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. Willing and able to comply with the study procedures and provide written informed consent to participate in the study
3. Schedule for a clinically indicated ERCP

Exclusion Criteria:

1. Potentially vulnerable subjects, including, but not limited to pregnant women
2. Subjects for whom endoscopic techniques are contraindicated
3. Subjects who are currently enrolled in another investigational study that would directly interfere with the current study, without prior written approval from the sponsor
4. Investigator discretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Number of patients complete the ERCP procedure | During the procedure
  Ability to complete the ERCP procedure for the intended indication(s) without crossing to reusable duodenoscope.
  It is also considered as Exalt D's ability if the clinical effect is the same per the investigator's judgement in case of an endoscope change (non-Exalt D).

SECONDARY OUTCOMES:
Endoscopist qualitative rating | During the procedure
  Endoscopist rating of the Exalt single-use duodenoscope compared to their past experience with marketed reusable duodenoscopes as it pertains to various design and performance related attributes. Besides those criteria similar to Exalt DScope 01 study, assessment in this study will include imaging quality (brightness, color, photometry), overall maneuverability and overall satisfaction, which will be rated from 1-10, where 1 is the worst and 10 is the best.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoshen Li, Principal Investigator — Boao Super Hospital

IPD SHARING:
Plan to Share IPD: Undecided